CLINICAL TRIAL: NCT05079620
Title: Antibiotic Prophylaxis in Critically Ill Patients After Suspected Aspiration
Brief Title: Early Antibiotics After Aspiration in ICU Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Under-enrollment
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Mark Metersky, Chief, Division of Pulmonary, Critical Care and Sleep Medicine, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-004-02
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Aspiration; Aspiration Pneumonia
Keywords: ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration; Pneumonia, Ventilator-Associated | interventions — Ceftriaxone; Amoxicillin-Potassium Clavulanate Combination; Cefepime; Vancomycin; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotics (Experimental): 5 days of empiric antibiotics selected from a guideline-appropriate regimen. Alternate agents may be selected by the treating team if allergies or other patient factors mandate, but are still recommended for a 5 day course. Supportive care including oxygen and ventilation can be offered ad libitum.
  Options include ceftriaxone, Augmentin, cefepime, vancomycin, levofloxacin.
  Interventions: Drug: Ceftriaxone; Drug: Amoxicillin clavulanic acid; Drug: Cefepime; Drug: Vancomycin; Drug: Levofloxacin
- Control (No Intervention): No initial antibiotic therapy unless clinical picture changes or worsens. Supportive care including oxygen and ventilation can be offered ad libitum.

INTERVENTIONS:
Drug: Ceftriaxone — If there is low risk for P. aeruginosa and/or methicillin-resistant staphylococcus aureus (MRSA), as deemed by the treating team: Ceftriaxone 2 g IV, every 24 hours for 5 days
  Arms: Antibiotics
Drug: Amoxicillin clavulanic acid — At any point after 24 hours, clinicians may (but are not required to) transition stable patients on ceftriaxone to the oral agent Amoxicillin + clavulanate (Augmentin) 875 mg PO or per feeding tube, twice daily for the remainder of 5 days
  Other Names: Augmentin
  Arms: Antibiotics
Drug: Cefepime — If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Cefepime 2 g IV, every 8 hours for 5 days, plus vancomycin
  Arms: Antibiotics
Drug: Vancomycin — If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Vancomycin IV, dosed by trough or AUC/MIC (area under the curve/minimum inhibitory concentration) monitoring for 5 days, plus cefepime. Order nasal MRSA swab and consider discontinuing vancomycin if MRSA swab is negative.
  Arms: Antibiotics
Drug: Levofloxacin — At any point after 24 hours, clinicians may (but are not required to) transition stable patients on cefepime to levofloxacin PO or per feeding tube, 750 mg every 24 hours for the remainder of 5 days
  Arms: Antibiotics

SUMMARY:
The purpose of this study is to evaluate the use of early antibiotics in ICU patients who appear to have aspirated, to help determine whether this improves outcomes by reducing the later incidence of pneumonia and other negative consequences.

DETAILED DESCRIPTION:
ICU patients with signs of aspiration on imaging and a clinical history supportive of aspiration, but with no clear signs of infectious pneumonia, will be randomized to receive either 5 days of empiric antibiotics or supportive care only. They will be followed for 30 days with a primary outcome of ICU length-of-stay and various secondary outcomes including mortality, ventilator days, and antibiotic days.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU within the last 24 hours, or with a witnessed aspiration event in the last 24 hours while in the ICU
* Radiographic findings on chest x-ray or CT deemed by the treating ICU team to be consistent with aspiration (e.g. dependent infiltrates or intraluminal airway debris)
* Clinical history consistent with possible aspiration (e.g. cardiac arrest, found unconscious, or with a witnessed aspiration event).

Exclusion Criteria:

* Already received 3 or more doses of any antibiotic since hospital presentation, unless the last dose was greater than 1 week before enrollment
* Requires antibiotic therapy for the treatment of other infections
* Patient "comfort measures only" at time of screening
* Currently participating in other trials using investigational drugs or interventions
* Currently pregnant
* Currently a prisoner
* The consenting party (patient or their legally authorized representative) is unable to understand or read English at a fifth-grade level.
* 2 or more of the following are present at the time of screening:
* White blood cell count: ≥ 11.0
* Temperature ≥ 38.0C (100.4F)
* Purulent secretions
* S/F (pulse oximetry saturation to FiO2) ratio ≤ 215

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Oto, Study Director — UConn Health, Adult Critical Care
Locations (1):
- UConn Health, John Dempsey Hospital, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dragan V, Wei Y, Elligsen M, Kiss A, Walker SAN, Leis JA. Prophylactic Antimicrobial Therapy for Acute Aspiration Pneumonitis. Clin Infect Dis. 2018 Aug 1;67(4):513-518. doi: 10.1093/cid/ciy120. PMID 29438467
- [Background] Acquarolo A, Urli T, Perone G, Giannotti C, Candiani A, Latronico N. Antibiotic prophylaxis of early onset pneumonia in critically ill comatose patients. A randomized study. Intensive Care Med. 2005 Apr;31(4):510-6. doi: 10.1007/s00134-005-2585-5. Epub 2005 Mar 8. PMID 15754197
- [Background] DiBardino DM, Wunderink RG. Aspiration pneumonia: a review of modern trends. J Crit Care. 2015 Feb;30(1):40-8. doi: 10.1016/j.jcrc.2014.07.011. Epub 2014 Jul 22. PMID 25129577
- [Background] El-Solh AA, Pietrantoni C, Bhat A, Aquilina AT, Okada M, Grover V, Gifford N. Microbiology of severe aspiration pneumonia in institutionalized elderly. Am J Respir Crit Care Med. 2003 Jun 15;167(12):1650-4. doi: 10.1164/rccm.200212-1543OC. Epub 2003 Apr 10. PMID 12689848
- [Background] Francois B, Cariou A, Clere-Jehl R, Dequin PF, Renon-Carron F, Daix T, Guitton C, Deye N, Legriel S, Plantefeve G, Quenot JP, Desachy A, Kamel T, Bedon-Carte S, Diehl JL, Chudeau N, Karam E, Durand-Zaleski I, Giraudeau B, Vignon P, Le Gouge A; CRICS-TRIGGERSEP Network and the ANTHARTIC Study Group. Prevention of Early Ventilator-Associated Pneumonia after Cardiac Arrest. N Engl J Med. 2019 Nov 7;381(19):1831-1842. doi: 10.1056/NEJMoa1812379. PMID 31693806
- [Background] Lascarrou JB, Lissonde F, Le Thuaut A, Bachoumas K, Colin G, Henry Lagarrigue M, Vinatier I, Fiancette M, Lacherade JC, Yehia A, Joret A, Lebert C, Bourdon S, Martin Lefevre L, Reignier J. Antibiotic Therapy in Comatose Mechanically Ventilated Patients Following Aspiration: Differentiating Pneumonia From Pneumonitis. Crit Care Med. 2017 Aug;45(8):1268-1275. doi: 10.1097/CCM.0000000000002525. PMID 28594680
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Marik PE. Aspiration syndromes: aspiration pneumonia and pneumonitis. Hosp Pract (1995). 2010 Feb;38(1):35-42. doi: 10.3810/hp.2010.02.276. PMID 20469622
- [Background] Marik PE, Careau P. The role of anaerobes in patients with ventilator-associated pneumonia and aspiration pneumonia: a prospective study. Chest. 1999 Jan;115(1):178-83. doi: 10.1378/chest.115.1.178. PMID 9925081
- [Background] Rebuck JA, Rasmussen JR, Olsen KM. Clinical aspiration-related practice patterns in the intensive care unit: a physician survey. Crit Care Med. 2001 Dec;29(12):2239-44. doi: 10.1097/00003246-200112000-00001. PMID 11801813
- [Background] Sirvent JM, Torres A, El-Ebiary M, Castro P, de Batlle J, Bonet A. Protective effect of intravenously administered cefuroxime against nosocomial pneumonia in patients with structural coma. Am J Respir Crit Care Med. 1997 May;155(5):1729-34. doi: 10.1164/ajrccm.155.5.9154884.
- [Background] Valles J, Peredo R, Burgueno MJ, Rodrigues de Freitas AP, Millan S, Espasa M, Martin-Loeches I, Ferrer R, Suarez D, Artigas A. Efficacy of single-dose antibiotic against early-onset pneumonia in comatose patients who are ventilated. Chest. 2013 May;143(5):1219-1225. doi: 10.1378/chest.12-1361. PMID 23715136

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiotics: 5 days of empiric antibiotics selected from a guideline-appropriate regimen. Alternate agents may be selected by the treating team if allergies or other patient factors mandate, but are still recommended for a 5 day course. Supportive care including oxygen and ventilation can be offered ad libitum.
  Options include ceftriaxone, Augmentin, cefepime, vancomycin, levofloxacin.
  Ceftriaxone: If there is low risk for P. aeruginosa and/or methicillin-resistant staphylococcus aureus (MRSA), as deemed by the treating team: Ceftriaxone 2 g IV, every 24 hours for 5 days
  Amoxicillin clavulanic acid: At any point after 24 hours, clinicians may (but are not required to) transition stable patients on ceftriaxone to the oral agent Amoxicillin + clavulanate (Augmentin) 875 mg PO or per feeding tube, twice daily for the remainder of 5 days
  Cefepime: If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Cefepime 2 g IV, every 8 hours for 5 days, plus vancomycin
  Vancomycin: If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Vancomycin IV, dosed by trough or AUC/MIC (AUC/MIC) monitoring for 5 days, plus cefepime. Order nasal MRSA swab and consider discontinuing vancomycin if negative.
  Levofloxacin: At any point after 24 hr, clinicians may (but are not required to) transition stable patients on cefepime to levofloxacin PO or per feeding tube, 750 mg q 24 hours for the remainder of 5 days
Period: Overall Study
Arm/Group | Antibiotics | Control
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Antibiotics: 5 days of empiric antibiotics selected from a guideline-appropriate regimen. Alternate agents may be selected by the treating team if allergies or other patient factors mandate, but are still recommended for a 5 day course. Supportive care including oxygen and ventilation can be offered ad libitum.
  Options include ceftriaxone, Augmentin, cefepime, vancomycin, levofloxacin.
  Ceftriaxone: If there is low risk for P. aeruginosa and/or methicillin-resistant staphylococcus aureus (MRSA), as deemed by the treating team: Ceftriaxone 2 g IV, every 24 hours for 5 days
  Amoxicillin clavulanic acid: At any point after 24 hours, clinicians may (but are not required to) transition stable patients on ceftriaxone to the oral agent Amoxicillin + clavulanate (Augmentin) 875 mg PO or per feeding tube, twice daily for the remainder of 5 days
  Cefepime: If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Cefepime 2 g IV, every 8 hours for 5 days, plus vancomycin
  Vancomycin: If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Vancomycin IV, dosed by trough or AUC/MIC (AUC/MIC) monitoring for 5 days, plus cefepime. Order nasal MRSA swab and consider discontinuing vancomycin if negative.
  Levofloxacin: At any point after 24 hours, clinicians may (but are not required to) transition stable patients on cefepime to levofloxacin PO or per feeding tube, 750 mg every 24 hours for the remainder of 5 days
- Total: Total of all reporting groups
Arm/Group | Antibiotics | Control | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (4.2) | 76.7 (19.4) | 72.8 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Intubated prior to enrollment [Count of Participants; unit: Participants] | 1 | 1 | 2
Chronic tracheostomy [Count of Participants; unit: Participants] | 0 | 0 | 0
Current steroid use at time of enrollment [Count of Participants; unit: Participants] | 0 | 1 | 1
Witnessed aspiration event, prior to admission [Count of Participants; unit: Participants] | 0 | 1 | 1
Days between hospital admission and enrollment [Mean (Standard Deviation); unit: days] | 0 (0) | 2 (3.5) | 1.2 (2.7)
Pneumonia diagnosed prior to enrollment [Count of Participants; unit: Participants] | 0 | 0 | 0
Positive serum ethanol at time of admission [Count of Participants; unit: Participants] | 0 | 0 | 0
Positive sputum culture prior to enrollment [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: ICU-free Days
Description: Number of days not spent in the ICU, between date of admission and 30 days afterwards. Death or discharge can both reduce this measure.
Time Frame: From admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Mean (Standard Deviation); unit: days
Groups:
- Antibiotics: 5 days of empiric antibiotics selected from a guideline-appropriate regimen. Alternate agents may be selected by the treating team if allergies or other patient factors mandate, but are still recommended for a 5 day course. Supportive care including oxygen and ventilation can be offered ad libitum.
  Options include ceftriaxone, Augmentin, cefepime, vancomycin, levofloxacin.
  Ceftriaxone: If there is low risk for P. aeruginosa and/or methicillin-resistant staphylococcus aureus (MRSA), as deemed by the treating team: Ceftriaxone 2 g IV, every 24 hours for 5 days
  Amoxicillin clavulanic acid: At any point after 24 hours, clinicians may (but are not required to) transition stable patients on ceftriaxone to the oral agent Amoxicillin + clavulanate (Augmentin) 875 mg PO or per feeding tube, twice daily for the remainder of 5 days
  Cefepime: If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Cefepime 2 g IV, every 8 hours for 5 days, plus vancomycin
  Vancomycin: If there is significant risk of P. aeruginosa and/or MRSA as deemed by the treating team: Vancomycin IV, dosed by trough or AUC/MIC monitoring for 5 days, plus cefepime. Order nasal MRSA swab and consider discontinuing vancomycin if negative.
  Levofloxacin: At any point after 24 hours, clinicians may transition stable patients on cefepime to levofloxacin PO or per feeding tube, 750 mg q24 hours for the remainder of 5 days
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
days | 14 (14.1) | 18.7 (16.1)

2. Secondary Outcome: Ventilator-free Days
Description: Number of days without any mechanical ventilation, between date of admission and 30 days afterwards. Death, discharge, or mechanical ventilation can both reduce this measure.
Time Frame: From admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
days | 19 (15.6) | 20 (17.3)

3. Secondary Outcome: Hospital-free Days
Description: Number of days not spent in the hospital, between date of admission and 30 days afterwards. Death or discharge can both reduce this measure.
Time Frame: From admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
days | 9 (12.7) | 14.7 (13.7)

4. Secondary Outcome: Antibiotic-free Days
Description: Number of days without any antibiotics administered, between date of admission and 30 days afterwards. Death, discharge, or antibiotic use can all reduce this measure.
Time Frame: Days with no antibiotics from admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
days | 12 (17) | 14 (14.5)

5. Secondary Outcome: Number of Participants Intubated After Enrollment
Description: Yes/no
Time Frame: Between admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Who Underwent Tracheostomy After Enrollment
Description: Yes/no
Time Frame: Between admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

7. Secondary Outcome: Number of Participants Who Developed Pneumonia After Enrollment
Description: Yes/no, by criteria: 2 or more present simultaneously of temperature >38c, WBC >11k, S/F ratio <215, and purulent secretions
Time Frame: Between admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 1 | 1

8. Secondary Outcome: Days Before Developing Pneumonia Criteria
Description: By criteria: 2 or more present simultaneously of temperature >38c, WBC >11k, S/F ratio <215, and purulent secretions
Time Frame: Between admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 1 | 1
days | 0 (0) | 0 (0)

9. Secondary Outcome: Number of Participants Prescribed Additional Antibiotics After Enrollment
Description: Yes/no. Excluding prophylactic antibiotics and excluding perioperative prophylactic antibiotics.
Time Frame: Between admission to 30 days, death, or hospital discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 1 | 2

10. Secondary Outcome: Number of Participants With a Positive Sputum Culture With a Presumed Pathogen
Description: Yes/no
Time Frame: Between enrollment and 30 days, death, or hospital discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

11. Secondary Outcome: Number of Participants With Any Positive Culture With an Organism Resistant to Prophylactic Antibiotics
Description: Yes/no
Time Frame: Between admission and 30 days, death, or hospital discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With a Positive C. Difficile Stool Toxin Assay After Enrollment
Description: Yes/no
Time Frame: Between enrollment and 30 days, death, or hospital discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

13. Secondary Outcome: Number of Participants With a Temperature >38 Centigrade on Day 3
Description: Yes/no
Time Frame: Day 3 after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

14. Secondary Outcome: Number of Participants With a White Blood Cell Count >11k on Day 3
Description: Yes/no
Time Frame: Day 3 after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 1 | 2

15. Secondary Outcome: Number of Participants With Arterial Oxygen Saturation / Fraction of Inspired Oxygen (S/F) <215 on Day 3
Description: Yes/no
Time Frame: Day 3 after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

16. Secondary Outcome: Number of Participants With Purulent Secretions on Day 3
Description: Yes/no
Time Frame: Day 3 after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

17. Secondary Outcome: 30 Day Mortality
Description: Death within 30 days from enrollment
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotics | Control
Number analyzed (Participants) | 2 | 3
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 30 days from enrollment
Arm/Group | Antibiotics | Control
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT05079620/Prot_SAP_001.pdf